CLINICAL TRIAL: NCT06106113
Title: Pharmacokinetics and Safety of GST-HG171 Tablets in Subjects With Impaired and Normal Liver Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Fujian Akeylink Biotechnology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GST-HG171-I-02
Record Dates: First submitted 2022-12-29; First posted 2023-10-30 (Actual); Last update posted 2023-10-30 (Actual); Status verified 2022-12

CONDITIONS: COVID-19 Pneumonia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mild hepatic impairment (Other): 150 mg GST-HG171
  Interventions: Drug: GST-HG171 Tablets
- Moderate hepatic impairment (Other): 150 mg GST-HG171
  Interventions: Drug: GST-HG171 Tablets
- healthy subjects with normal hepatic function (Other): 150 mg GST-HG171
  Interventions: Drug: GST-HG171 Tablets

INTERVENTIONS:
Drug: GST-HG171 Tablets — 150mg GST-HG171 Tablets

SUMMARY:
This si a single-center, non-randomized, open, parallel, single-dose trial was designed to evaluate the safety and pharmacokinetic characteristics of GST-HG171 tablets in subjects with impaired liver function.

ELIGIBILITY:
Inclusion Criteria:

All subjects are required to meet all of the following conditions

1. Voluntarily sign informed consent prior to the start of activities related to this study, be able to understand the procedures and methods of this study, and be willing to strictly follow the clinical trial protocol to complete this study;
2. Subjects (including their partners) are willing to have no family planning and voluntarily take highly effective contraception within 6 months after the last study drug administration;
3. Age range from 18 to 65 (including both ends) on the date of signing the informed consent, both male and female;
4. Male subjects should weigh no less than 50 kg and female subjects should weigh no less than 45 kg; Body mass index (BMI) 18-32 kg/m2 (including both ends);
5. Creatinine clearance (calculated by Cockcroft-Gault formula) ≥60 mL/min;

   Subjects with normal liver function should also meet all of the following conditions:
6. The following demographic matching criteria must be met during screening:

   1. Body weight was matched with that of the group with liver function impairment, with an average of ±10 kg;
   2. Age matching was performed between the group with liver function impairment, the mean was ±10 years old;
   3. Gender matching was performed with liver function impairment group, and the mean was ±1 case;

   Subjects with impaired liver function should also meet all of the following conditions:
7. Chronic liver injury caused by primary liver diseases (such as hepatitis B, hepatitis C, autoimmune hepatitis, alcoholic liver disease, etc.), liver insufficiency patients with Child-Pugh grade A or B;
8. Cirrhosis was clinically diagnosed;
9. Stable medication regimen for liver dysfunction, complications and other concomitant diseases for at least 14 days prior to taking the study drug, and no adjustment of medication (including type, dosage or frequency of medication) is required; Or have not used drugs;

Exclusion Criteria:

Subjects meeting any of the following exclusion criteria will not be enrolled in this study

1. Allergic constitution, including severe drug allergy or history of drug allergy, known allergy to the study drug or any component of the study drug;
2. During the screening period, electrocardiogram showed QTc interphase (QTcF) >470 msec for males and >480 msec for females (corrected according to Fridericia's standard);
3. A history of dysphagia or any gastrointestinal disorder affecting drug absorption, including frequent nausea or vomiting due to any etiology;
4. Patients with severe infection, trauma, gastrointestinal surgery or other major surgical operations within 4 weeks before screening;
5. Those who had been vaccinated within 14 days prior to screening or planned to be vaccinated during the study period;
6. Those who donated blood or lost more than 200 mL of blood within 3 months prior to screening, or intended to donate blood during the trial or within 1 month after the trial;
7. A strong or medium acting inducer or inhibitor of CYP3A enzyme, a strong P-glycoprotein (P-gp) inhibitor or inducer used within 1 month before screening;
8. D1 had taken a special diet (including dragon fruit, mango, grapefruit, and/or xanthine diet, chocolate) and/or consumed excessive amounts of tea, coffee, grapefruit/grapefruit juice and/or caffeinated beverages (more than 8 cups of 200 mL per cup per day on average) in the 2 weeks prior to administration;
9. Binge drinkers in the 3 months preceding screening, i.e. those who consume more than 14 units of alcohol per week (1 unit = 360 mL beer, or 45 mL spirits with 40% alcohol by volume, or 150 mL wine) or those who test positive for alcohol; Smokers who smoked at least 10 cigarettes a day in the 3 months before screening;
10. Those who have a history of drug use, or drug abuse, or test positive for drug abuse;
11. Pregnant or lactating women or women of childbearing age who have tested positive for pregnancy;
12. Patients who cannot tolerate venipunction or have a history of fainting needle and fainting blood;
13. Those not suitable for inclusion for other reasons;

    Subjects with normal liver function should be excluded if they meet any of the following exclusion criteria:
14. History of liver injury;
15. Have been or are currently suffering from any clinically serious disease such as circulatory system, endocrine system, nervous system, digestive system, respiratory system, hematology, immunology, psychiatric and metabolic abnormalities, or any other disease that may interfere with the test results;
16. Physical examination, vital signs, laboratory examination, 12-lead electrocardiogram, abdominal color ultrasound and other abnormalities were judged by researchers to have clinical significance;
17. Hepatitis B surface antigen, hepatitis C antibody or hepatitis C core antigen, HIV antigen/antibody or syphilis antibody positive for any index;
18. Study the use of any prescription, over-the-counter, Chinese herbal or supplement within 14 days prior to drug administration;
19. Use of other clinical trial drugs within 3 months prior to screening or plan to participate in other clinical trials.

    Subjects with liver function impairment who meet any of the following exclusion criteria shall be excluded:
20. The subject has any of the following conditions: drug-induced liver injury; History of liver transplantation; In addition, patients with cirrhosis that is considered to be complicated by the following complications, including but not limited to liver failure, hepatic encephalopathy, hepatocellular carcinoma, esophageal varicose hemorrhage, etc.;
21. The laboratory test results during screening were consistent with any of the following: (a) alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >10×ULN; (b) neutrophil absolute value (NE#) <0.75×109/L; (c) Hemoglobin (HGB) <60 g/L; (d) alpha-fetoprotein (AFP) >100 ng/mL;
22. HIV antigen/antibody screening positive; If syphilis antibody is positive, rapid plasma rereaction hormone test (RPR) should be added. If RPR is positive at the same time, it should be excluded.
23. In addition to the primary liver disease itself, those who have had or currently suffered from other serious systemic organ diseases, including but not limited to gastrointestinal, respiratory, kidney, nervous, blood, endocrine, tumor, immune, psychiatric or cardiovascular and cerebrovascular diseases, or abnormal clinical laboratory tests have clinical significance, and are judged by the study doctor to be unfit to participate in this study;
24. Participants who used other clinical trials within 1 month prior to screening or planned to participate in other clinical trials during the study period.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2022-12-15 (Actual); Primary Completion 2023-02-06 (Actual); Study Completion 2023-05-30 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration (Cmax) for GST-HG171 | Day 1 at 0 (pre-dose) ,0.25 ,0.5 ,0.75 ,1 ,1.25 ,1.5 ,2 ,3 ,4 ,6 ,8 ,12 ,24 and 48 hours post-dose
  Maximum observed plasma GST-HG171 concentration.

SECONDARY OUTCOMES:
AEs | up to Day 7
  To evaluate the safety and tolerability of GST-HG171 tablets after a single oral administration in subjects with mild and moderate liver impairment and normal liver function

CONTACTS AND LOCATIONS:
Locations (1):
- The first hospital of Jilin University, Changchun, Jilin, China

REFERENCES:
- [Derived] Zhou J, Zhang H, Chen H, Zhang G, Mao J, Zhang T, Tang Y, Yan W, Li C, Ding Y, Jin Q. Pharmacokinetics and safety of GST-HG171, a novel 3CL protease inhibitor, in Chinese subjects with impaired and normal liver function. Antimicrob Agents Chemother. 2024 Aug 7;68(8):e0053924. doi: 10.1128/aac.00539-24. Epub 2024 Jul 11. PMID 38990016